CLINICAL TRIAL: NCT05833022
Title: Patient Characteristics and Treatment Patterns From Early Crizanlizumab Use in Real-world Setting: Preliminary Analysis From Select Sickle Cell Centers
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CSEG101AUS16
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This was a retrospective cohort study using secondary data from member sites of the National Alliance of Sickle Cell Centers (NASCC) with at least five patients who initiated crizanlizumab. Patients who were prescribed crizanlizumab were included in the cohort.

ELIGIBILITY:
Inclusion criteria:

* Any patient with diagnosis of SCD based on high-performance liquid chromatography (HPLC) or hemoglobin electrophoresis at treating institution
* Treatment order for crizanlizumab; Index date was defined as the date for the first crizanlizumab treatment
* At least 12 months of available electronic medical record (EMR) data pre-index date (baseline)
* Patients must have received at least one dose of crizanlizumab
* For inclusion in pre/post analysis of effectiveness, patients must have received at least 6 doses of medication. The rates could be annualized if total post-index time was <12 months.

Exclusion criteria:

None specified

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who received sickle cell disease treatment (use of hydroxyurea, l-glutamine, chronic transfusion therapy, and voxelotor) prior to treatment with crizanlizumab | Up to 12 months
Percentage of patients who received sickle cell disease treatment (use of hydroxyurea, l-glutamine, chronic transfusion therapy, and voxelotor) during treatment with crizanlizumab | Up to 12 months

SECONDARY OUTCOMES:
Number of patients who discontinued treatment with crizanlizumab | Up to 24 months
Number of doses of crizanlizumab for patients who discontinued treatment with crizanlizumab | Up to 24 months
Reasons for early discontinuation of crizanlizumab treatment | Up to 24 months
Number of sickle cell disease (SCD)-related hospitalizations | Up to 24 months
Number of SCD-related emergency department (ED) visits | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (11):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Cristiana Care, Wilmington, Delaware
  - All Children's Hospital, St. Petersburg, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University of St. Louis, St Louis, Missouri
  - Beth Israel Hospital, East Hanover, New Jersey
  - Montefiore, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University Hospital at Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Texas (Houston), Houston, Texas